CLINICAL TRIAL: NCT01532219
Title: Internet-delivered Psychodynamic Therapy for Depression and Anxiety Disorders: A Randomized Controlled Trial
Brief Title: Internet-delivered Psychodynamic Therapy for Depression and Anxiety Disorders
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor of Clinical Psychology, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-DEPANX2012-APT
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-delivered Psychodynamic Treatment (Experimental): Participants in the experimental condition will receive 8 text-modules delivered as guided self-help, via the Internet. The intervention lasts for 10 weeks and includes weekly contacts with a therapist via a secure online environment similar to e-mail. The treatment is a short-term psychodynamic treatment psychodynamic treatment.
  Interventions: Behavioral: Internet-delivered Psychodynamic Treatment
- Internet-delivered structured support (Active Comparator): Participants in the active control condition will receive a structured support treatment via the Internet. The intervention lasts for 10 weeks and includes weekly contacts with a therapist via a secure online environment similar to e-mail.
  Interventions: Behavioral: Internet-delivered structured support

INTERVENTIONS:
Behavioral: Internet-delivered Psychodynamic Treatment — Ten weeks of guided self-help + therapist contact, via the Internet.
  Arms: Internet-delivered Psychodynamic Treatment
Behavioral: Internet-delivered structured support — Ten weeks of therapist contact, via the Internet.
  Arms: Internet-delivered structured support

SUMMARY:
The overall aim of this study is to develop and test a psychodynamic Internet-delivered psychological treatment for patients with major depression and/or anxiety disorders and compare its efficacy to an active control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder, Panic Disorder, Social Anxiety Disorder, Generalized Anxiety disorder, Depressive Disorder NOS or Anxiety Disorder NOS
* 10 or higher on the PHQ-9 or on the GAD-7 at pre-treatment

Exclusion Criteria:

* Primary diagnosis of Obsessive Compulsive Disorder or Post-traumatic Stress Disorder
* Severe psychiatric condition (e.g. psychosis or bipolar disorder)
* Alcohol abuse (more than 16 on the AUDIT)
* Suicidal (measured in diagnostic interview)
* Changed medication during the last three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
9-item Patient Health Questionnaire Depression Scale (PHQ-9) | Two weeks before the treatment starts
7-item Patient Health Questionnaire Generalized Anxiety Disorder Scale (GAD-7) | Two weeks before the treatment starts
9-item Patient Health Questionnaire Depression Scale (PHQ-9) | At treatment start (0 weeks)
7-item Patient Health Questionnaire Generalized Anxiety Disorder Scale (GAD-7) | At treatment start (0 weeks)
9-item Patient Health Questionnaire Depression Scale (PHQ-9) | At treatment termination (10 weeks)
7-item Patient Health Questionnaire Generalized Anxiety Disorder Scale (GAD-7) | At treatment termination (10 weeks)
9-item Patient Health Questionnaire Depression Scale (PHQ-9) | At treatment follow-up (7 months)
7-item Patient Health Questionnaire Generalized Anxiety Disorder Scale (GAD-7) | At treatment follow-up (7 months)

SECONDARY OUTCOMES:
Emotional Processing Scale (EPS-25) | Two weeks before the treatment starts
Emotional Processing Scale (EPS-25) | At treatment start (0 weeks)
Emotional Processing Scale (EPS-25) | At treatment termination (10 weeks)
Five Facets of Mindfulness Questionnaire (FFMQ) | Two weeks before the treatment starts
Five Facets of Mindfulness Questionnaire (FFMQ) | At treatment start (0 weeks)
Five Facets of Mindfulness Questionnaire (FFMQ) | At treatment termination (10 weeks)
Emotional Processing Scale (EPS-25) | At treatment follow-up (7 months)
Five Facets of Mindfulness Questionnaire (FFMQ) | At treatment follow-up (7 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University, Department of Behavioral Sciences and Learning, Linköping, Sweden